CLINICAL TRIAL: NCT04240444
Title: A Prospective, Multicenter, Randomized Controlled Clinical Trial to Assess the Safety and Efficacy of SeQuent® SCB Balloon in the Treatment of Patients With Coronary Arteries In-stent Restenosis Compared SeQuent® Please Neo
Brief Title: Sirolimus-Coated Balloon Versus Paclitaxel-Coated Balloon for the Treatment of Coronary In-Stent Restenosis
Acronym: SIBLINT ISR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B. Braun Medical International Trading Company Ltd. (Industry)
Collaborators: CCRF Inc., Beijing, China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAG-G-H-1905
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease; In Stent Restenosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SeQuent® SCB (Experimental): patients will receive sirolimus (rapamycin)-coated balloon (SeQuent® SCB)
  Interventions: Device: drug-coated balloon Catheter
- SeQuent® Please Neo (Active Comparator): patients will receive SeQuent® Please Neo balloon
  Interventions: Device: drug-coated balloon Catheter

INTERVENTIONS:
Device: drug-coated balloon Catheter — All eligible subjects will be assigned randomly to study group or control group, receive PTCA.

SUMMARY:
This is a prospective, multicenter, randomized controlled clinical trial, which plans to enroll 260 subjects.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized (1:1) controlled clinical trial, which plans to enroll 260 subjects. The aim of study is to assess the safety and efficacy of SeQuent® SCB in the treatment of in-stent restenosis in coronary arteries.

All eligible subjects with ISR lesion in coronary will be randomly assigned to receive SeQuent® SCB (study group) or receive SeQuent® Please Neo (control group) balloon treatment. All subjects will be scheduled to clinical follow up at 30 days, 6 months, 9 months and 12 months after index procedure and will be scheduled to receive the angiography at 9 months after index procedure. The primary endpoint was segment late luminal loss at 9 months after index procedure.

ELIGIBILITY:
Inclusion Criteria:

* General criteria

  1. Patient ≥18 years of age.
  2. Stable angina pectoris or unstable angina pectoris (acute coronary syndrome), prior myocardial infarction or proven asymptomatic myocardial ischemia.
  3. Patients are eligible for any type of coronary revascularization.
  4. Patients agree to receive angiography follow-up at 9 months after index procedure.
  5. Patients agree to receive clinical follow-up at 30 days, 6months, 9 months and 1years after index procedure.
  6. Patients are able to understand the purpose of the study and will comply with the study protocol. The patient is willing to sign informed consent form and understand the risks and benefits described in the informed consent form.
* lesion related

  1. Up to 2 ISR lesions which found by angiography (diameter stenosis ≥70% or ≥ 50% with evidence of ischemia) or functional examination (e.g. FFR<0.8 IVUS<4mm2) will be treated, target segment includes news lesions within 5mm of the stent margin.
  2. Up to 2 drug coated balloons (SeQuent® Please Neo or SeQuent® SCB) will be used in the study, with 1 drug coated balloon per lesion.
  3. ISR (including bare stents, inert and active drug eluting stents) : Mehran type I, II and III stenosis; The reference vessel diameter of target lesions ranges from 2.5mm to 4.0mm (visual), and the length of each lesion are≤ 34mm (visual).
  4. Other de novo lesions needing treatment must be >10mm away from the target lesion.

Exclusion Criteria:

* General criteria

  1. Patients with myocardial infarction within 1 week before index procedure.
  2. Patients with takayasu arteritis.
  3. Patients with severe renal failure, whose Creatinine >2.0 mg/dL (177 mol/L).
  4. LVEF<30%.
  5. Hb before procedure <10 g/dL.
  6. Patients with Coagulation disorder, platelet count <100,000/mm3.
  7. Patients with cardiogenic shock.
  8. Patients with diseases who require cytostatic or radiotherapy.
  9. Patients who are known to be allergic or contraindicated to aspirin, heparin, clopidogrel, rapamycin, ticagrelor, tirofiban, paclitaxel, or iopromide , or who are allergic to contrast agents and cannot be medically prevented, or who are on cilostazol anticoagulants.
  10. Patients with bleeding conditions, or with conditions that increase the risk of bleeding, such as gastrointestinal ulcers, which may be restricted or prohibited from anticoagulant therapy or the use of anticoagulant drugs.
  11. Gestational women who were pregnant before receiving treatment with the study device or who planned to be pregnant during the study , and did not use effective contraception until (including) follow-up at 12 months postoperatively; Female patients during lactation.
  12. Patients with a life expectancy less than 1 year.
  13. Patients who are participating in any other clinical trial.
  14. Investigator considered the patients ineligible due to any reasons.
* lesion related

  1. There are more than 3 lesions to be treated (including non-target lesions to be treated), and there are more than 2 lesions to be treated in each coronary artery.
  2. There will be more than 5 stents implanted in coronary artery after intervention (including previous and current PCI).
  3. After pre-dilatation of target lesion, there will be residual stenosis of target lesion >30% or TIMI blood flow < grade 3, and/ dissections NHLBI grade C,D,E,F.
  4. The ISR lesion has been treated in past 6 months.
  5. The target lesion is tortuous, severely calcified, angular, and the DCB is expected to be impassable.
  6. Target lesion contains thrombosis.
  7. Target or non-target lesion(s) located in left main.
  8. Patients with previous CABG.
  9. Patients with lesions requiring intervention treatment in 3 vessels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
In-segment late loss | at 9 months after index procedure
  In-segment late loss(LLL) is defined as the difference between the MLD immediately after the procedure and the MLD at 9-month follow-up angiography after index procedure. MLDs are measured by QCA.

SECONDARY OUTCOMES:
The success rate of intervention treatment | 1-3 days
  including device success, lesion success and clinical success
Binary restenosis rate of target lesion | 9 months after index procedure
  A diameter stenosis of > 50% at the previously treated lesion site, including the originally treated site plus the adjacent vascular segments 5 mm , proximal and 5 mm distal to the site . Percent diameter stenosis was defined as [1(MLD/reference vessel diameter)]100.
Target lesion failure (TLF) rate | 30 days, 6 months, 9 moths, 12 months after index procedure
  The composite of ischemia-driven revascularization of the target lesion, MI related to the target vessel, or cardiac death related to the target vessel
PoCE | 30 days, 6 months, 9 moths, 12 months after index procedure
  a composite of all death, MI and any revascularization
ARC-defined stent thrombosis | 30 days, 6 months, 9 moths, 12 months after index procedure
  timing (acute, subacute, late and very late stent thrombosis); relationship (definite, probable and possible stent thrombosis)

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, academician, Principal Investigator — The General Hospital of Northern Theater Command
Locations (16):
- China (16):
  - Anhui Provincal Hospital, Hefei, Anhui
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - Ruijin Hospital，Shanghai Jiaotong University，School of medicine, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Liu H, Li Y, Fu G, An J, Chen S, Zhong Z, Liu B, Qiu C, Ma L, Cong H, Li H, Tong Q, He B, Jin Z, Zhang J, Yuan H, Qiu M, Zhang R, Han Y. Sirolimus- vs Paclitaxel-Coated Balloon for the Treatment of Coronary In-Stent Restenosis: The SIBLINT-ISR Randomized Trial. JACC Cardiovasc Interv. 2025 Apr 28;18(8):963-971. doi: 10.1016/j.jcin.2024.12.024. Epub 2025 Feb 19. PMID 39985511